CLINICAL TRIAL: NCT02740439
Title: Investigating the Effects of Avocado Intake on Metabolism and Cognition: A Systems Approach
Brief Title: Persea Americana for Total Health (PATH ) Study
Acronym: PATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16277
Record Dates: First submitted 2016-04-11; First posted 2016-04-15 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Obesity, Abdominal; Insulin Resistance; Insulin Sensitivity
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Meal (Experimental): Intervention meals will contain 1 large avocado and be consumed daily for 12 weeks.
  Interventions: Other: Avocado
- Control Meal (Placebo Comparator): Control meals will be isocaloric to the intervention meals but without avocado. They will also be consumed daily for 12 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Avocado — The intervention meals will contain 1 large avocado.
  Arms: Intervention Meal
Other: Control — The control meals will be isocaloric to the intervention meals but will not contain avocado.
  Arms: Control Meal

SUMMARY:
The proposed work will investigate the effects of avocados on abdominal obesity and glycemic control among overweight/obese adults.

DETAILED DESCRIPTION:
The proposed work will investigate the effects of avocados on abdominal obesity and glycemic control among overweight/obese adults. Further, changes in GI microbiota composition and cognitive function will be assessed to comprehensively understand systemic benefits of avocado consumption on gut and brain function. This research study has two aims: 1) To determine the effects of regular avocado intake on metabolic syndrome risk factors, specifically, abdominal obesity and glycemic control, among overweight and obese adults; and 2) to investigate the implications of avocado intake on measures of GI microbiota composition and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Between the ages of 25-45 years at the time of consent
* Body mass index ≥27.5kg/m2
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision).
* Ability to drop-off fecal sample within 15 minutes of defecation

Exclusion Criteria:

* Current pregnancy or lactation
* Tobacco use
* Avocado allergy or intolerance
* Food allergies, lactose intolerance
* Latex allergy
* Prior diagnosis of metabolic and gastrointestinal disease (cardiovascular disease and type 1 or type 2 diabetes, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.)
* Prior diagnosis of cognitive or physical disability, including ADHD, severe asthma, epilepsy, chronic kidney disease, and dependence upon a wheelchair/walking
* Use of any anti-psychotic, anti-depressant, anti-anxiety, or ADD/ADHD medications
* Use of medications that alter normal bowel function and metabolism (e.g., recent antibiotic use, laxatives, enemas, anti-diarrheal agents, narcotics, antacids, antispasmodics, diuretics, anticonvulsants).
* High BMI that is not representative of being overweight or obese (e.g. resistance trained individuals, football players)
* Prior malabsorptive bariatric surgery (i.e. gastric bypass, sleeve gastrectomy) or restrictive bariatric surgery (i.e. adjustable gastric band) within the past 2 years

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Abdominal obesity | Baseline, 4 weeks, 8 weeks, 12 weeks
  Changes to abdominal and whole body composition including visceral and subcutaneous adipose tissue will be estimated by DEXA.
Glycemic Control | Baseline, 4 weeks, 8 weeks,12 weeks
  Glycemic control will be assessed using oral glucose tolerance tests and hemoglobin A1c.
Insulin Resistance | Baseline, 4 weeks, 8 weeks, 12 weeks
  Insulin resistance will be evaluated using the Homeostasis Assessment Model (HOMA) index.
Insulin Sensitivity | Baseline, 12 weeks
  Insulin sensitivity will be assessed using the insulinogenic index, Stumvoll Metabolic Clearance Rate, Oral Glucose Insulin Sensitivity, and the Matsuda Index.

SECONDARY OUTCOMES:
Gastrointestinal Microbiota Composition and Short Chain Fatty Acids | Baseline, 4 weeks, 8 weeks, 12 weeks
  Microbial taxonomy will be assessed using high throughput sequencing and short chain fatty acids will be quantified using gas chromatography and mass spectrometry.
Cognitive Function | Baseline, 4 weeks, 8 weeks, 12 weeks
  Cognitive function will be evaluated using tasks that measure prefrontal cognitive control and hippocampal relational memory networks.
Retinal Lutein | Baseline, 4 weeks, 8 weeks, 12 weeks
  Retinal lutein will be assessed using Macular Pigment Optical Density.
Serum Lutein | Baseline, 12 weeks
  Serum lutein will be assessed using venous blood samples.
Blood Lipid Panel | Baseline, 12 weeks
  Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides will be assessed using venous blood samples.
Resting Energy Expenditure | Baseline, 12 weeks
  REE will be measured by indirect calorimetry.
Neuroelectric Assessment | Baseline, 4 weeks, 8 weeks, 12 weeks
  A Neuroelectric Assessment will be conducted during cognitive tasks using an Electroencephalogram (EEG) amplifier.
DNA Analyses | Baseline
  Genetic markers related to obesity and cognitive function will be assessed using blood samples to determine the mediating effects of genetics on changes related to study outcomes.
Dietary Intake | Baseline, 4 weeks, 8 weeks, 12 weeks
  Dietary intake will be evaluated using 7 day diet records at baseline, 4, 8, and 12 weeks and by NCI NHANES 30-day food frequency questionnaires at baseline and 12 weeks.
Sleep and Fatigue | Baseline, 12 weeks
  Sleep and fatigue will be evaluated using the Pittsburgh Sleep Quality Index
Physical Activity | Baseline, 12 weeks
  Physical activity will be measured over 7 day periods by a waist mounted accelerometer.
Blood Pressure | Baseline, 12 weeks
  Blood pressure will be measured using an automatic blood pressure cuff.
Liver Enzymes | Baseline, 12 weeks
  Liver enzymes will be assessed using venous blood samples.
Inflammatory Markers | Baseline, 12 weeks
  Markers of inflammation such as c-reactive protein (CRP) will be assessed using venous blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah D Holscher, PhD RD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois, Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Derived] Hughes RL, Pindus DM, Khan NA, Burd NA, Holscher HD. Associations between Accelerometer-Measured Physical Activity and Fecal Microbiota in Adults with Overweight and Obesity. Med Sci Sports Exerc. 2023 Apr 1;55(4):680-689. doi: 10.1249/MSS.0000000000003096. Epub 2022 Dec 22. PMID 36728974
- [Derived] Khan NA, Edwards CG, Thompson SV, Hannon BA, Burke SK, Walk ADM, Mackenzie RWA, Reeser GE, Fiese BH, Burd NA, Holscher HD. Avocado Consumption, Abdominal Adiposity, and Oral Glucose Tolerance Among Persons with Overweight and Obesity. J Nutr. 2021 Sep 4;151(9):2513-2521. doi: 10.1093/jn/nxab187. PMID 34191028
- [Derived] Thompson SV, Bailey MA, Taylor AM, Kaczmarek JL, Mysonhimer AR, Edwards CG, Reeser GE, Burd NA, Khan NA, Holscher HD. Avocado Consumption Alters Gastrointestinal Bacteria Abundance and Microbial Metabolite Concentrations among Adults with Overweight or Obesity: A Randomized Controlled Trial. J Nutr. 2021 Apr 8;151(4):753-762. doi: 10.1093/jn/nxaa219. PMID 32805028
- [Derived] Edwards CG, Walk AM, Thompson SV, Reeser GE, Erdman JW Jr, Burd NA, Holscher HD, Khan NA. Effects of 12-week avocado consumption on cognitive function among adults with overweight and obesity. Int J Psychophysiol. 2020 Feb;148:13-24. doi: 10.1016/j.ijpsycho.2019.12.006. Epub 2019 Dec 14. PMID 31846631
- [Derived] Jones AR, Robbs CM, Edwards CG, Walk AM, Thompson SV, Reeser GE, Holscher HD, Khan NA. Retinal Morphometric Markers of Crystallized and Fluid Intelligence Among Adults With Overweight and Obesity. Front Psychol. 2018 Dec 21;9:2650. doi: 10.3389/fpsyg.2018.02650. eCollection 2018. PMID 30622502